CLINICAL TRIAL: NCT02842840
Title: The Effectiveness of Multimodal Educational Intervention to Improve Adherence to Treatment Regimens in Older Stroke Patients: A Randomised Trial
Brief Title: The Effectiveness of Multimodal Educational Intervention to Improve Adherence to Treatment Regimens in Older Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Associate Professor of health psychology, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR.QUMS.REC.1394.350
Record Dates: First submitted 2016-04-12; First posted 2016-07-25 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Stroke; Medication Adherence; Older Adults
MeSH Terms: conditions — Stroke; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Patients based intervention (Experimental): A multifaceted intervention program will use to improve adherence and clinical outcomes in Stroke patients. This intervention focus on behavioral treatment in the patients.
  Interventions: Behavioral: Patient-based intervention
- Family based intervention (Experimental): Patients and their families will receive a series of educational/motivational interventions.
  Interventions: Behavioral: Family based intervention
- Routine counseling (Active Comparator): All participants of the study in both group receive the Standard Care. Usually, patients in clinics receive a one-time session of brief advice to use medications regularly lasting approximately 30 minutes and deliver by nurse or physician. Some issues rise in this short session including coexisting diseases, the history of drug use, current disease and advice about the health risks of irregular medication use.
  Interventions: Other: Routine counseling

INTERVENTIONS:
Behavioral: Patient-based intervention
  Arms: Patients based intervention
Behavioral: Family based intervention
  Arms: Family based intervention
Other: Routine counseling
  Arms: Routine counseling

SUMMARY:
Stroke is a major cause of morbidity and mortality, especially in low and middle income countries including Iran. Patients with recent stroke or TIA are at high risk for new vascular events. Several evidence based strategies in secondary prevention of stroke are available but frequently underused. The study is aimed to evaluate an intervention to improve patients with Stroke.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* able to give informed consent

Exclusion Criteria:

* recurrent stroke
* a diagnosis of subarachnoid haemorrhage
* significant impairments precluding participation - inability to give informed consent
* another condition likely to impact their participation in the trial (e.g. life-threatening condition other than cardiovascular disease)
* expected discharge to hospital/nursing home setting

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
changes in Patient-reported Adherence Medication Adherence Rating Scale | changes from baseline, 6 Months, 12 months and 18 months follow-up
  a self-report measure of adherence (Medication Adherence Report Scale [MARS-5]) will be used .
changes in blood pressure | changes from baseline, 6 Months, 12 months and 18 months follow-up
changes in low-density lipoprotein (LDL)-cholesterol level | changes from baseline, 6 Months, 12 months and 18 months follow-up

SECONDARY OUTCOMES:
Changes in intention to medication adherence | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in Action Plan | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The action plan is assessed by a self-reported questionnaire. it is used by the patients before, at baseline, six months, twelve months and eighteen months after the intervention
Changes in Coping Plan | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The coping plan is assessed by a self-reported questionnaire. It is used by the patients before, at baseline, six months, twelve months and eighteen months after the intervention
Changes in quality of life | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The Short Form (36) Health Survey is used to assess patient's quality of life
Changes in perceived behavioral control to medication adherence | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The perceived behavioral control to medication adherence is assessed through a self-report instrument
Changes in Self-monitoring to medication adherence | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The Self-monitoring to medication adherence is assessed through a self-report instrument
Changes in Illness Perceptions | changes from baseline, 6 Months, 12 months and 18 months follow-up
  the Brief Illness Perception. Questionnaire (Brief IPQ) is used to assess patient's illness representation

CONTACTS AND LOCATIONS:
Locations (3):
- Iran (3):
  - Department of Public Health, Qazvin University of Medical Sciences, Qazvin, Qazvin Province
  - Qazvin University of Medical Sciences, Qazvin, Qazvin Province
  - Outpatient Pediatric Clinic, Qazvin, Qazvin Province